CLINICAL TRIAL: NCT00529022
Title: Phase I Trial of Sequential Azacitidine and Valproic Acid Plus Carboplatin in the Treatment of Patients With Platinum Resistant Epithelial Ovarian Cancer
Brief Title: Azacitidine and Valproic Acid Plus Carboplatin in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0030
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Solid Tumors
Keywords: Advanced Cancer; Solid Tumors; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Azacitidine; 5-Azacitidine; 5-Aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Vidaza; Valproic Acid; Depakene; Carboplatin; Paraplatin
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Azacitidine; Valproic Acid; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine + Valproic Acid + Carboplatin (Experimental): Azacitidine 75 mg/m^2 subcutaneous injection or by vein daily for 5 Days. Valproic Acid 40 mg/kg by mouth daily for 7 days. Carboplatin area under the curve (AUC) 2 by vein on Days 3 and 10 over 60 Minutes.
  Interventions: Drug: Azacitidine; Drug: Valproic Acid; Drug: Carboplatin

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m^2 Subcutaneous Injection or by vein Daily for 5 Days.
  Other Names: 5-Azacitidine; 5-Aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: Valproic Acid — 40 mg/kg by mouth Daily for 7 days.
  Other Names: Depakene
Drug: Carboplatin — AUC 2 by vein on Days 3 and 10 over 60 Minutes.
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research study is to find out if giving azacitidine with valproic acid plus carboplatin can help control advanced cancer. The safety of this treatment will be studied as well. Researchers will also collect some extra blood samples for molecular marker studies (studies that may help researchers predict how participants respond to the combined therapy).

There were to be two phases of this study: a Phase 1 portion to find acceptable doses of the study drug combination, and a Phase 2 portion to study the response rates to the treatment schedule. The study did not proceed to the Phase 2 portion.

DETAILED DESCRIPTION:
The Study Drugs:

Researchers want to see if the combination of azacitidine, carboplatin, and valproic may work better together to control advanced cancer.

* Azacitidine is designed to activate ("turn on") certain genes in cancer cells whose job is to fight tumors, which may also make azacitidine work better with other anti-tumor drugs.
* Carboplatin is designed to block the growth of cancer cells by stopping cell division, which may cause the cells to die.
* Valproic acid is an anti-seizure medication that may also have cancer-fighting abilities. This drug may be able to activate tumor-fighting genes, causing cancer cells to die.

Phase 1 (Dose Escalation) and Phase 2 (Treatment):

Participants will be enrolled on Phase 1 of the study in groups of 3. Each group will receive a different combination of the study drugs. If the first group of 3 tolerates the study drug combination well, the next group of 3 will be enrolled, and their dose(s) of carboplatin and/or valproic acid will be higher than the last group. Each new group will get a higher dose of carboplatin and/or valproic acid. If 1 of the 3 participants has a serious side effect at a certain dose level, 3 more participants may be added at that dose level to check the safety of the combination. If no more participants at that dose level have serious side effects, the next dose level will be tested. However, if a second participant has a serious side effect, then the dose level before that one will be considered the "maximum tolerated dose" (MTD). Once the MTD is found, participants will be enrolled on Phase 2 of the study.

Participants enrolled on Phase 2 were to be given the MTD level of the study drug combination; however, study did not progress to Phase 2.

Participants on both phases were to have the same treatment schedule and study tests performed. The only difference between Phase 1 and Phase 2 was to be the dose level of the study drug combination being given.

Study Treatment:

If eligible, participants received the study treatment on a 28-day treatment cycle.

On Day 1 of each cycle, they receive an injection of azacitidine just under the skin or by vein over 30 minutes once a day for 5 days in a row.

On Day 3 and Day 10 of each cycle, they receive carboplatin by vein over 60 minutes.

On Days 5-11 of each cycle, they take valproic acid by mouth once a day with or without food.

On Day 12 of each cycle, they may receive an injection of NeulastaTM (pegfilgrastim) just under the skin, depending on whether the study doctor thinks it is needed to help boost your white blood cell count.

On Days 13-28 of each cycle, they have a "rest period" from the study drugs before beginning a new 28-day cycle of treatment.

Study Visits:

At certain time points, they have the following tests/procedure performed during study visits:

On Day 5 and Day 11 of Cycles 1-3, about 1 tablespoon of blood drawn before treatment for molecular marker studies. These tests will be performed to look for a link between genetic characteristics and response to the study drug treatment.

Within the last 72 hours (3 days) of each cycle, blood drawn (about 1 tablespoon) and urine collected for routine tests. After the start of each cycle, blood drawn (about 1 tablespoon) once weekly for routine tests.

Within 7 days before starting each new cycle, evaluation to see if you may be experiencing any side effects.

After the end of every 2 cycles (about every 8 weeks), an x-ray and either a CT scan or an MRI scan to re-evaluate the cancer.

Length of Study:

Participants will continue to receive treatment on this study, as long as the disease does not get worse and you do not experience any intolerable side effects.

End-of-Treatment Visit:

Once treatment has ended for any reason, participants will come back for an end-of-treatment visit to have the following tests/procedures performed:

* You will have a complete physical exam.
* You will have urine collected and blood drawn (about 1 tablespoon) for routine tests.
* You may have a CT scan or an MRI scan to remeasure and re-evaluate the cancer.

Up to 65 patients were eligible to take part in this study. All were to be enrolled at M. D. Anderson. Study halted after Phase 1 without progressing to second phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed diagnosis of advanced solid tumor (that has progressed following standard therapy or for whom, in the opinion of the investigator, no standard effective therapy is available) during the phase I study. Only patients who have platinum resistant epithelial carcinoma of the ovary, fallopian tube or primary peritoneal carcinoma are enrolled onto the phase 2 study, if progresses to phase 2. According to standard Gynecologic Oncology Group (GOG) criteria platinum resistant is defined to have had a disease-free interval of shorter than 6 months following platinum treatment.
2. Patient has measurable or evaluable disease by radiological imaging techniques with documented progression within 1 month before study entry or disease that has not responded to treatment. (Pleural effusions, ascites, osseous metastasis, elevation of tumor marker and lesions located in previously irradiated areas are not considered measurable).
3. Patient is willing to comply with study procedures to have blood collections for correlative studies.
4. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Patient must be informed of the investigational nature of this study and must sign and give written Internal Review Board (IRB) approved informed consent in accordance with institutional guidelines.
6. If patient is of child-bearing potential, she or he has agreed to practice an effective method of birth control during the study and up to 3 months after the last treatment.
7. Patient has adequate liver and renal function: serum albumin =/>3.0 g/dL; serum bilirubin =/<2.0 mg/dL; alanine aminotransferase (ALT) =/<3* upper limit of normal (uln); and serum creatinine =/< 2.0 mg/dL or a calculated creatinine clearance of at least 40 ml/min.
8. Patient has adequate bone marrow reserve. Absolute neutrophil count (ANC) =/>1,500/ul, Platelet count =/>100,000/ul, and Hemoglobin =/>9.0g/dL.

Exclusion Criteria:

1. Any concurrent chemotherapy.
2. Underlying medical condition that might be aggravated by treatment or that cannot be controlled, such as active uncontrolled serious infection and cardiac dysfunction.
3. Medical and psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk.
4. Known hypersensitivity to azacitidine, valproic acid, carboplatin or their analogs.
5. Failure to recover from any prior surgery within 4 weeks of study entry.
6. Pregnant or lactating.
7. Any treatment specific for tumor control within 3 weeks of dosing with study drugs (within 2 weeks if given weekly or within 6 weeks for nitrosoureas or mitomycin C) or failure to recover from the toxic effect of any of these therapies prior to study entry. Any investigational drug within 30 days of first day of dosing.
8. Any signs of intestinal obstruction interfering with nutrition or oral intake.
9. History of central nervous system (CNS) metastasis unless the patient has had surgery or radiation, and does not require oral or intravenous corticosteroids or anticonvulsants.
10. Advanced malignant hepatic tumors that are defined as the total hepatic metastases more than 25% of hepatic parenchyma.
11. History of high dose chemotherapy for ovarian cancer in phase 2 of the study, if Phase 2 of study needed. High dose chemotherapy is defined as the intensity and/or the density of a chemotherapeutic agent that are beyond standard of care for ovarian cancer treatment.
12. History of prior malignancy except for adequately treated carcinoma in situ of the uterine cervix, basal cell or squamous cell skin cancer, or other cancer for which the patient has been disease free for at least two years in phase 2 study, if Phase 2 of study needed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Response Rate | 8 weeks
  Assessment of tumor response by palpation, plain x-ray, MRI, or CT scan to be obtained after the first cycle and the every 2 cycles after that (8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Falchook, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Falchook GS, Fu S, Naing A, Hong DS, Hu W, Moulder S, Wheler JJ, Sood AK, Bustinza-Linares E, Parkhurst KL, Kurzrock R. Methylation and histone deacetylase inhibition in combination with platinum treatment in patients with advanced malignancies. Invest New Drugs. 2013 Oct;31(5):1192-200. doi: 10.1007/s10637-013-0003-3. Epub 2013 Aug 2. PMID 23907406
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org